CLINICAL TRIAL: NCT00066950
Title: Prevention Management Model for Early Childhood Caries
Brief Title: Prevention Management Model for Early Childhood Caries (MAYA Project)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Ysidro Health Center (Other); University of California, San Diego (Other); San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NIDCR-14251
Record Dates: First submitted 2003-08-07; First posted 2003-08-08 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Dental Caries
Keywords: Early childhood caries
MeSH Terms: conditions — Dental Caries | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling Only (No Intervention): Oral Health Counseling Only
- CHX+Counseling (caregiver) + FV (child) (Experimental): Oral Health Counseling plus Chlorhexidine for caregiver plus fluoride varnish every 6 months from 12mo to 30mo of age for child
  Interventions: Drug: Chlorhexidine gluconate; Device: Fluoride Varnish

INTERVENTIONS:
Drug: Chlorhexidine gluconate — 0.5oz chlorhexidine gluconate 0.12% solution mouth rinse twice daily for 14 days then no rinse for 14 days, repeated for 3 months
  Other Names: Peridex® OMNII Oral Pharmaceuticals
  Arms: CHX+Counseling (caregiver) + FV (child)
Device: Fluoride Varnish — 0.25ml FV every 6 months from age 12 to 30 months
  Other Names: CavityShield® OMNII Oral Pharmaceuticals
  Arms: CHX+Counseling (caregiver) + FV (child)

SUMMARY:
The purpose of this study is to determine whether dental disease patterns and transmissable bacteria that are known to cause a severe form of dental decay in young children can be reduced or eliminated by treating mothers and their young infants early on with Chlorhexidine and fluoride varnish applications, respectively as part of a comprehensive Prevention Management Model.

DETAILED DESCRIPTION:
The primary aim is to evaluate two programs, a minimal intervention program and a moderate intensity program, for preventing Early Childhood Caries. A four-year randomized clinical trial will be conducted specifically to: 1) Assess demographic and behavioral factors as predictors of ECC and the relationship between three-year post-intervention behavioral changes from baseline measures with disease outcomes; 2) Compare the efficacy for the prevention of ECC in two groups - the minimal intervention group (Group 1) receiving counseling alone, with the moderate intensity group (Group 2) receiving a) counseling and a therapeutic four-month regimen of Chlorhexidine rinse for new mothers and b) fluoride varnish applications for their infants and toddlers starting at twelve months of age and continuing to age 30 months; 3) Assess baseline salivary microbiological markers as predictors of ECC in the infants of women in both groups and the relationship between three-year post-intervention salivary markers and changes from baseline measures with disease outcomes; 4) Assess the impact of a caries-preventive model in lowering the salivary mutans streptococci level in post-partum women, and subsequently, in inhibiting the growth of these bacteria in their young children, delaying the infectious process.

The long term objectives are to build upon our understanding of caries risk factors, to assess the effectiveness of a prevention management model, to improve access to preventive oral health services and information for low-income pregnant women and their young children, and to reduce oral health disparities in a border population (U.S. - Mexico Border near San Diego Bay Area) at high risk for dental disease.

ELIGIBILITY:
"Inclusion Criteria"

* Some evidence of geographic stability in South San Diego Bay Area
* Planning on remaining in area approximately 3 years after birth of child
* Must be able to provide consent in English or Spanish
* Must be registered patients at San Ysidro Health Center in the prenatal program
* Must be experiencing a normal pregnancy

"Exclusion Criteria"

* Diabetes, anemia, placenta previa, seizure disorders, GDM, evidence of chromosomal disorders, Polyhydramnios, Thrombophlebitis, or RH-negative status
* Vaginal bleeding, premature uterine contractions, viral or bacterial infections, diabetes, pregnant with twins or multiple births expected
* Previous pregnancy complications where hospitalization was required

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 361 (Actual)
Dates: Start 2003-03; Primary Completion 2005-07 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Caries Incidence and Caries Index | 4 year
  Caries Incidence (number of participants who developed caries during the study) and the number of decayed or filled tooth surfaces (dfs) index.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Ramos-Gomez, DDS,MS, MPH, Principal Investigator — University of California, Los Angeles; Stuart A Gansky, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- San Ysidro Health Center, San Ysidro, California, United States

REFERENCES:
- [Result] Ramos-Gomez F, Chung LH, Gonzalez Beristain R, Santo W, Jue B, Weintraub J, Gansky S. Recruiting and retaining pregnant women from a community health center at the US-Mexico border for the Mothers and Youth Access clinical trial. Clin Trials. 2008;5(4):336-46. doi: 10.1177/1740774508093980. PMID 18697848
- [Result] Ramos-Gomez FJ, Gansky SA, Featherstone JD, Jue B, Gonzalez-Beristain R, Santo W, Martinez E, Weintraub JA. Mother and youth access (MAYA) maternal chlorhexidine, counselling and paediatric fluoride varnish randomized clinical trial to prevent early childhood caries. Int J Paediatr Dent. 2012 May;22(3):169-79. doi: 10.1111/j.1365-263X.2011.01188.x. Epub 2011 Oct 17. PMID 21999806
- [Result] Chaffee BW, Gansky SA, Weintraub JA, Featherstone JD, Ramos-Gomez FJ. Maternal oral bacterial levels predict early childhood caries development. J Dent Res. 2014 Mar;93(3):238-44. doi: 10.1177/0022034513517713. Epub 2013 Dec 19. PMID 24356441